CLINICAL TRIAL: NCT00093457
Title: A Phase II Study Of BAY 43-9006 (NSC 724772; CTEP IND# 69,896) In Patients With Hormone Refractory Prostate Cancer
Brief Title: Sorafenib in Treating Patients With Metastatic or Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I167; CAN-NCIC-IND167 (Other: PDQ); CDR0000387987 (Other: PDQ)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: sorafenib tosylate — BAY 43-9006 given orally at 400 mg BID in a 28 day cycle

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase II trial is studying the effectiveness of sorafenib in treating patients who have metastatic or recurrent prostate cancer that has not responded to previous hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of sorafenib, as measured by prostate-specific antigen response, in patients with metastatic or recurrent hormone-refractory adenocarcinoma of the prostate.

Secondary

* Determine the objective response rate and duration of response in patients treated with this drug.
* Determine the tolerability and toxicity of this drug in these patients.
* Determine time to treatment failure and overall survival in patients treated with this drug.
* Explore the relationship between measures of ras/raf pathway activation (pERK) and response to treatment in these patients.

OUTLINE: This is a non-randomized, multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks after going off study treatment and then periodically for survival. Patients with stable or responding disease, when they go off study treatment, are followed every 3 months until relapse or progression.

PROJECTED ACCRUAL: Approximately 15-25 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Metastatic or recurrent disease
* No curative standard therapy exists
* Hormone-refractory disease

  * Evidence of prostate-specific antigen (PSA) progression during androgen ablation therapy, including medical or surgical castration

    * Documented PSA progression after completion of prior peripheral anti-androgens

      * At least a 25% increase (≥ 5 ng/mL) over a reference value PSA with 2 consecutive rising PSAs taken ≥ 1 week apart
    * Castrate level of testosterone ≤ 1.7 nmol/L for patients on medical androgen ablation

      * Patients receiving luteinizing hormone-releasing hormone agonist therapy must continue this treatment during study participation
* PSA ≥ 10 ng/mL at the time of study entry
* Primary tumor tissue (paraffin embedded) must be available for immunohistochemistry
* Minimal symptomatic disease

  * No requirement for morphine or equivalent dose > 30 mg/day to control pain
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No evidence of bleeding diathesis

Hepatic

* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal

Renal

* Serum creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No myocardial infarction within the past 6 months
* No congestive heart failure
* No unstable angina
* No active cardiomyopathy
* No unstable ventricular arrhythmia
* No uncontrolled hypertension

Other

* No serious infection
* No active peptic ulcer disease
* No upper gastrointestinal or other condition that would preclude study compliance with oral medication
* No uncontrolled psychotic disorder
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to sorafenib or other study agents
* No other serious illness or medical condition that would preclude study participation
* No other malignancy within the past 5 years except adequately treated non-melanoma skin cancer or other curatively treated solid tumor

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Concurrent prophylactic filgrastim (G-CSF), sargramostim (GM-CSF), or other growth factors allowed for the management of adverse events only

Chemotherapy

* No prior chemotherapy
* No other prior cytotoxic chemotherapy

Endocrine therapy

* See Disease Characteristics
* Concurrent steroids allowed provided there has been no increase in steroid requirements within the past 4 weeks AND no increase in dose is planned

Radiotherapy

* At least 4 weeks since prior external-beam radiotherapy except low-dose non-myelosuppressive radiotherapy
* Concurrent low-dose non-myelosuppressive palliative radiotherapy allowed

Surgery

* Not specified

Other

* No prior investigational anticancer agents
* No concurrent therapeutic anticoagulation

  * Concurrent prophylactic low-dose warfarin for venous or arterial access devices allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy
* No other concurrent investigational therapy
* No concurrent grapefruit juice
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-08-10 (Actual); Primary Completion 2006-09-28 (Actual); Study Completion 2011-01-18 (Actual)

PRIMARY OUTCOMES:
Prostate-specific antigen response and/or progression | 2 years

SECONDARY OUTCOMES:
Objective response and/or progression | 2 years
Tolerability and toxicity | 2 years
Time to treatment failure and overall patient survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kim N. Chi, MD, Study Chair — British Columbia Cancer Agency
Locations (7):
- Canada (7):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chi KN, Ellard SL, Hotte SJ, Czaykowski P, Moore M, Ruether JD, Schell AJ, Taylor S, Hansen C, Gauthier I, Walsh W, Seymour L. A phase II study of sorafenib in patients with chemo-naive castration-resistant prostate cancer. Ann Oncol. 2008 Apr;19(4):746-51. doi: 10.1093/annonc/mdm554. Epub 2007 Dec 3. PMID 18056648